CLINICAL TRIAL: NCT00967434
Title: Short Term Atorvastatin Regime for Vasculopathic Surgical (STAR-VaS) Patients Study
Brief Title: Statin Drugs to Prevent Complications During Surgery
Acronym: STAR-VaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006832-01H
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Inflammation; Myocardial Infarction; Myocardial Ischemia
Keywords: infarction; ischemia; surgery; perioperative; statins
MeSH Terms: conditions — Inflammation; Myocardial Infarction; Myocardial Ischemia; Infarction; Ischemia | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A- atorvastatin in pre and postop (Active Comparator): Atorvastatin 80 mg administered daily for at least 7 preoperative days, 80 mg on day of surgery and 80 mg daily for up to 7 postoperative days.
  Interventions: Drug: Atorvastatin
- Group B- Atorvastatin postop (Active Comparator): Placebo administered for up to 7 preoperative days, atorvastatin 80 mg administered on day of surgery and daily for up to 7 postoperative days.
  Interventions: Drug: Atorvastatin
- Group C- Placebo (Placebo Comparator): Patients receive placebo daily for up 7 preoperative days, placebo on day of surgery and placebo daily for up to 7 postoperative days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — atorvastatin 80 mg daily for at least 7 preoperative days atorvastatin 80 mg on day of surgery atorvastatin 80 mg daily for up to 7 postoperative days
  Other Names: lipitor
  Arms: Group A- atorvastatin in pre and postop
Drug: Atorvastatin — Daily placebo on the preoperative days atorvastatin 80 mg on day of surgery atorvastatin 80 mg daily for up to 7 postoperative days
  Other Names: Lipitor
  Arms: Group B- Atorvastatin postop
Drug: Placebo — Daily placebo in preoperative period Placebo on day of surgery Daily placebo for up to 7 postoperative days
  Arms: Group C- Placebo

SUMMARY:
Patients undergoing non-cardiac surgery frequently experience perioperative cardiac complications that may be due to excess inflammatory reactions. Lipid lowering drugs called HMG-CoA reductase inhibitors or statins, have anti-inflammatory effects. Although favourable evidence suggests these drugs could also prevent perioperative cardiac complications, definitive evidence of anti-inflammatory effects and benefit is lacking. The purpose of this study to measure the impact of a atorvastatin on patients undergoing surgery. It will attempt to determine the speed of drug effect as measured by the impact the drug has on the levels of the inflammatory mediator called C-reactive protein after surgery. It is hypothesized that the perioperative use of atorvastatin will safely reduce the postoperative rise in CRP levels at 48 hours after elective vascular surgery. This effect, would then translate into a reduction of adverse perioperative complications including reduction in postoperative myocardial ischemia episodes (as measured through Holter monitoring).

DETAILED DESCRIPTION:
Despite modern improvements in operative care, non-cardiac surgery is still associated with significant and costly cardiac complications. The incidence of major perioperative cardiac events varies, ranging from 1% in unselected populations to 15% or more in vascular surgical patients. An estimated 2 million North Americans yearly experience a perioperative cardiac event with an associated mortality of 30-50% and financial burden of over 20 billion dollars. Best evidence suggests that medical optimization is the preferred strategy to reduce the risks. There exists favorable physiologic evidence and promising clinical observations that statin drugs may prevent perioperative complications. We propose a randomized controlled trial to evaluate short-term atorvastatin versus placebo on inflammatory changes and myocardial ischemia in patients undergoing high-risk non-cardiac surgery.

The traditional belief on the etiology of perioperative myocardial events has been that supply-demand discrepancies due to hypotension or hypoxia compromise cardiac oxygen delivery thus resulting in myocardial ischemia and infarction are in dispute. Therapies that target supply-demand imbalance, including perioperative beta-blockers, have been disappointing. Emerging evidence now suggests that most perioperative cardiac events are similar to non-operative events where rupture of coronary plaques and thrombosis are central to the development of acute coronary events. Key elements to plaque rupture are inflammation and endothelial dysfunction. Elevated inflammatory markers, particularly C-reactive protein is associated with adverse cardiac events. Drugs known as statins offer benefits beyond their traditional improvement of lipid levels. Statins have so-called pleiotropic effects that include anti-inflammatory, endothelial function changes and plaque stabilization. Atorvastatin, a statin with a good safety profile, is particularly effective at improving inflammatory levels and decreasing cardiac events including death.

Perioperatively, elevated C-reactive protein levels after surgery are associated with perioperative complications including cardiac events. Thus, strategies to control perioperative inflammation may reduce complications. Retrospective studies and small prospective studies suggest that statins would reduce perioperative complications but definitive evidence is lacking. Questions regarding dose and timing of dosing is unclear. Likewise, little is proven on the potential pathophysiology of atorvastatin on reducing perioperative myocardial events. Our hypothesis is that atorvastatin use will reduce the postoperative rise in CRP levels at 48 hours.

Eligible non-cardiac surgical patients will be randomized into 3 groups with 3 stages of treatment; namely stage 1 (preoperative period up to 7 days), stage 2 (immediate preoperative), and stage 3 (first 7 postoperative days). Group A will receive atorvastatin in all 3 stages. Group B receives placebo in stage 1 but atorvastatin stages 2 and 3. Group C receives placebo in all 3 stages. Atorvastatin dose in all cases will be 80 mg. C-reactive protein and lipid levels assess statin effects. Safety is assessed by liver enzymes and CK levels. Myocardial events assessed by troponin T, ECG and Holter monitoring. Follow-up at 6 months will be done.

ELIGIBILITY:
Inclusion Criteria:

* elective high-risk surgery defined by use of the POISE criteria
* over 45 years of age

Exclusion Criteria:

* lack of informed consent
* contraindication to statin (i.e. liver insufficiency or cirrhosis, active muscular disorder or myopathy, or previous adverse reaction to statin)
* pregnant
* enrolled in another conflicting study
* previously enrolled in STAR VaS
* presently using a statin drug

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
C-reactive protein levels at 48 hours postoperatively | 48 hours

SECONDARY OUTCOMES:
perioperative myocardial ischemia as detected by Holter monitoring | 48 hours
perioperative myocardial injury as measured by troponin levels | up to 7 postoperative days
liver enzyme levels | up to 7 postoperative days
myopathy as assessed by CK levels | up to 7 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: David T Neilipovitz, MD, Principal Investigator — The Ottawa Hospital; Greg L Bryson, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Neilipovitz DT, Bryson GL, Taljaard M. STAR VaS--Short Term Atorvastatin Regime for Vasculopathic Subjects: a randomized placebo-controlled trial evaluating perioperative atorvastatin therapy in noncardiac surgery. Can J Anaesth. 2012 Jun;59(6):527-37. doi: 10.1007/s12630-012-9702-z. Epub 2012 Apr 13. PMID 22528165